CLINICAL TRIAL: NCT06744998
Title: Hemopatch Implication After Axillary Dissection for Breast Cancer: a Randomized Clinical Study
Brief Title: Hemopatch Implication After Axillary Dissection for Breast Cancer
Acronym: BreastPatch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: L2-249
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Primary breast cancer; Axillary dissection; Axillary seroma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective monocentric controlled randomized surgical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemopatch® group (Experimental): Hemopatch® application after axillary dissection
  Interventions: Device: Hemopatch® (Baxter)
- No Hemopatch® group (No Intervention): No Hemopatch® application after axillary dissection

INTERVENTIONS:
Device: Hemopatch® (Baxter) — HEMOPATCH® is an absorbable collagen pad intended for sealing and hemostasis
  Arms: Hemopatch® group

SUMMARY:
Aim of this randomized study is to assess the value of a different haemostatic sealant, the Hemopatch®, in axillary lymph node dissection (ALND) to reduce the incidence of seroma and seroma-related complications.

DETAILED DESCRIPTION:
With the de-escalation of axillary lymph node dissection (ALND) to sentinel lymph node biopsy as a surgical procedure staging in breast cancer (BC), the physical and psychological morbidity has been improved significantly. However, ALND is still considered in a relevant number of BC patients as treatment for controlling locoregional axillary disease, and these patients present still important complications related to ALND, such as neuropathy, limitation of shoulder movement, arm lymphedema, and most commonly seroma evolution.

Multiple surgical devices with the intent to improve sealing of lymphatic and blood vessels have demonstrated contrasting results in the incidence of seroma formation after ALND and are no utilized routinary. Non-surgical devices, such as chemical medications, sealing small vessels by stimulating collagen and fibrinogen syntheses, also could improve to sealing of the lymphatic vessels. Additionally, fibrin glue-coated collagen patches and fibrin glue application to the surgical cavity were already tested in ALND patients with contrasting benefit in term of seroma prevention. Unfortunately, none of these studies provided a good solution to eliminate or reduce the incidence of seroma after ALND in BC treatment.

Aim of this randomized study is to assess the value of a different haemostatic sealant, the Hemopatch®, in axillary lymph node dissection (ALND) to reduce the incidence of seroma and seroma-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary breast cancer
* Mastectomy or breast conserving surgery
* Patients eligible for axillary dissection
* Male or female
* Any age
* Previous (or not) neoadjuvant treatments
* Any breast histotypes

Exclusion Criteria:

* Previous axillary surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Axillary seroma evaluation | 1 week
  Measure of drain output (in cc) in one week

SECONDARY OUTCOMES:
Hospital access evaluation | 1 month
  Total number of hospital accesses per patient within one month post-surgery
Drain duration evaluation | 1 month
  Time until drain removal (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Corso, MD, PhD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy